CLINICAL TRIAL: NCT00281827
Title: Phase II Trial of Neoadjuvant Therapy With Carboplatin and Gemcitabine With Thalidomide in Patients With Stage II and IIIA Non-Small Cell Lung Cancer
Brief Title: Carboplatin, Gemcitabine, and Thalidomide in Patients Undergoing Surgery for Stage II or III Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to drug unavailability
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002LS013; LILLY-X-382 (Other: Eli Lilly); 0202M17981 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Results first posted 2009-12-03 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Lung Cancer
Keywords: adenocarcinoma of the lung; squamous cell lung cancer; large cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Gemcitabine; Thalidomide; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Chemotherapy treatment (carboplatin, gemcitabine and thalidomide) every 21 days for 3 courses.
  Interventions: Drug: carboplatin; Drug: gemcitabine hydrochloride; Drug: thalidomide; Procedure: conventional surgery

INTERVENTIONS:
Drug: carboplatin — Day 1 of Cycles 1, 2 and 3 - intravenously (IV) 30 minutes (Area Under the Curve = 5.5)
  Other Names: PARAPLATIN
Drug: gemcitabine hydrochloride — Days 1 and 8 of Cycles 1, 2 and 3 - 30 minute IV, 1000 mg/m2.
  Other Names: Gemzar
Drug: thalidomide — Oral administration: Cycle 1 - Day 1 50 mg, Day 2 100 mg, Day 3 150 mg, Day 4 and continuing until end of study treatment 200 mg.
  Other Names: Thalidomid
Procedure: conventional surgery — Resection - between 2 and 6 weeks following last dose of chemotherapy.
  Other Names: Surgery; Resection

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Thalidomide may stop the growth of tumor cells by blocking blood flow to the tumor. Giving carboplatin and gemcitabine together with thalidomide before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well giving carboplatin and gemcitabine together with thalidomide works in treating patients who are undergoing surgery for stage II or stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the complete and partial response rates in patients with stage II or IIIA non-small cell lung cancer treated with neoadjuvant carboplatin, gemcitabine hydrochloride, and thalidomide.

Secondary

* Determine, preliminarily, the mechanism of action and activity of thalidomide against lung cancer.
* Determine the 1-year and 2-year survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine the operative mortality of patients treated with this regimen.

OUTLINE: This is a pilot study.

Patients receive carboplatin intravenously (IV) over 30 minutes on day 1, gemcitabine hydrochloride IV over 30 minutes on days 1 and 8, and oral thalidomide once daily on days 1-21. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Within 2-6 weeks after the completion of chemotherapy, patients with resectable tumors undergo surgical resection.

After completion of study treatment, patients are followed every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC), including any of the following histologic subtypes:

  * Squamous cell carcinoma
  * Adenocarcinoma
  * Large cell undifferentiated carcinoma
* Stage II or IIIA disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral Computerized Axial Tomography (CT) scan
* No tumor involving the superior sulcus (e.g., Pancoast tumor)
* Karnofsky performance status 70-100%
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 2 mg/dL
* Bilirubin < 2 mg/dL
* Aspartate aminotransferase (AST) < 3 times upper limit of normal

Exclusion Criteria:

* Pregnant or nursing

  * No nursing during and for ≥ 4 weeks after completion of study treatment
* Positive pregnancy test
* Fertile female patients must use 2 effective methods of contraception 4 weeks before, during, and for 4 weeks after completion of study treatment
* Fertile male patients must use effective barrier contraception during and for 4 weeks after completion of study treatment
* Blood, sperm, or ova donation during study treatment
* Post obstructive pneumonia
* Other serious infection or medical illness that would preclude study participation
* Other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or other malignancy that is unlikely to affect survival for the next 3 years
* Less than 5 years since prior resection of lung disease
* Prior systemic chemotherapy or radiotherapy for non-small cell lung cancer (NSCLC)
* Other concurrent chemotherapy or radiotherapy
* Concurrent hormonal therapy or immunotherapy
* Other concurrent anticancer therapy
* Other concurrent investigational agents
* Concurrent participation in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2002-05; Primary Completion 2008-03 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arkadiusz Dudek, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (3):
- United States (3):
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 3 participating study centers.
Groups:
- Intent-to-Treat: Patients receiving at least one dose of each study drug (carboplatin, gemcitabine and thalidomide).
Period: Overall Study
Arm/Group | Intent-to-Treat
Started | 22
Completed | 22 (All patients received 3 cycles of therapy; 2 did not receive all 3 thalidomide cycles)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intent-to-Treat
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 53 [32 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Reporting Clinical Response
Description: Objective clinical response measuring using tumor assessments: Complete Response (CR) = disappearance of all target and non-target lesions and normalization of tumor marker level, if applicable. Pathological Complete Response (PCR) = No viable tumor cells in specimen determined by light microscopy. Partial Response (PR) = at least 30% decrease in the sum of longest diameter of target lesions from baseline. Progressive Disease (PD) = at least 20% increase in the sum of longest diameters of target lesions from baseline or new lesions. Stable Disease (SD) = Neither PR or PD.
Time Frame: At end of 3 -21 day cycles of treatment
Population: 2 of 22 patients did not receive all 3 drugs for all 3 cycles - only 20 patients achieved this and are thereby included here in the evaluable population analysis.
Measure: Number; unit: Participants
Groups:
- Evaluable Patients: Patients receiving 3 complete cycles of treatment (all 3 drugs over 3 - 21 day time periods).
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 20
Participants
  Complete Response | 0
  Pathological Complete Response | 0
  Partial Response | 14
  Stable Disease | 4
  Progressive Disease | 2

2. Secondary Outcome: Number of Patients Disease-free at 1 Year
Description: Calculated from date of enrollment to date of recurrence or death, whichever came first
Time Frame: 1 year
Population: Calculated from study entry date to date of recurrence or date of death, whichever came first.
Measure: Number; unit: Participants
Arm/Group | Intent-to-Treat
Number analyzed (Participants) | 22
Participants | 14 [1.117 to 2.954]

3. Secondary Outcome: Number of Patients Disease-free at 2 Years
Description: Calculated from date of enrollment to date of recurrence or death, whichever came first
Time Frame: 2 Years
Measure: Number; unit: Participants
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 22
Participants | 8

4. Secondary Outcome: Number of Patients Alive at 1 Year (Survival)
Description: Participants who were alive at one year from date of enrollment .
Time Frame: 12 Months
Population: Calculated from date of first date of enrollment.
Measure: Number; unit: Participants
Arm/Group | Intent-to-Treat
Number analyzed (Participants) | 22
Participants | 21

5. Secondary Outcome: Number of Patients Alive at 2 Years (Survival)
Description: Participants who were alive at 2 years from date of enrollment.
Time Frame: 24 Months
Population: Calculated from date of first date of enrollment to date of death.
Measure: Number; unit: Participants
Arm/Group | Intent-to-Treat
Number analyzed (Participants) | 22
Participants | 16

6. Secondary Outcome: Number of Patients Alive at 56 Months (End of Study)
Description: Patients alive from date of enrollment to date of death or censored at date of last contact (Overall Survival).
Time Frame: Up to 56 months
Population: Calculated from study entry date to date of death or censored at date of last contact.
Measure: Number; unit: Participants
Arm/Group | Intent-to-Treat
Number analyzed (Participants) | 22
Participants | 8 [1.938 to NA]

ADVERSE EVENTS:
Time Frame: Events were collected from Day 1 of study through 30 days post last treatment.
Arm/Group | Intent-to-Treat
Serious Adverse Events (participants affected / at risk) | 1/19
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intent-to-Treat (N=19)
Carotid stenosis (Vascular disorders) | 1 (1) — Visceral arterial ischemia (non-myocardial), not related to thalidomide.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intent-to-Treat (N=22)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 7 (10)
Anorexia (Gastrointestinal disorders) | 3 (3)
Anxiety (Nervous system disorders) | 2 (4)
Appetite loss (Gastrointestinal disorders) | 2 (2)
Breast, left, soreness (Musculoskeletal and connective tissue disorders) | 1 (1)
Cold sensation (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 17 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Depression (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Dizziness (Nervous system disorders) | 7 (8)
Double vision (Eye disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3)
Dyseugsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) — Due to fall
Edema, extremity (Blood and lymphatic system disorders) | 5 (7)
Edema, facial (Skin and subcutaneous tissue disorders) | 1 (2)
Elevated transaminase (Metabolism and nutrition disorders) | 1 (1)
Epistaxis/nosebleed (Vascular disorders) | 1 (1)
Erythemia intravenous arm site (Skin and subcutaneous tissue disorders) | 1 (1)
Fainting spell (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 13 (22)
Fever episode (General disorders) | 2 (2)
Flu-like symptoms (General disorders) | 4 (5)
General body aches (General disorders) | 1 (1)
General malaise (General disorders) | 1 (1)
Headaches, intermittent (Nervous system disorders) | 3 (3)
Hearing loss diagnosis (Ear and labyrinth disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 2 (2)
Hemoptisis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness, loss of voice (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hot flashes (Endocrine disorders) | 1 (1)
Hyperpigmentation of skin on nose (Skin and subcutaneous tissue disorders) | 1 (1)
Hypersensitive to cold (General disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Irritable (Nervous system disorders) | 1 (1)
Itching/pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Leg aches (Musculoskeletal and connective tissue disorders) | 1 (1)
Moodiness (Nervous system disorders) | 1 (1)
Mouth lesions (bumps) (Skin and subcutaneous tissue disorders) | 1 (1)
Mouth/tongue sensitivity (Gastrointestinal disorders) | 2 (3)
Mucositis (Gastrointestinal disorders) | 3 (4)
Muscle aches (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 14 (18)
Neuropathy, lower extremities (Nervous system disorders) | 4 (5)
Neutropenia (Blood and lymphatic system disorders) | 12 (14)
Nocturia (Renal and urinary disorders) | 1 (1)
Numbness, jaw and cheek (Nervous system disorders) | 1 (1)
Numbness, right side (Nervous system disorders) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Pain, PIC line site (Skin and subcutaneous tissue disorders) | 1 (1)
Pain, ankle (Gastrointestinal disorders) | 1 (1) — Twisted ankle, tripped and fell
Pain, central chest (General disorders) | 1 (1)
Pain, ear (General disorders) | 1 (1)
Pain, jaw (General disorders) | 1 (1)
Pain, low back (General disorders) | 2 (2)
Pain, rib (General disorders) | 1 (1)
Pain/cramps, abdominal (General disorders) | 1 (1)
Rash, body (Skin and subcutaneous tissue disorders) | 10 (12)
Rash, facial (Skin and subcutaneous tissue disorders) | 3 (4)
Rash, peripheral (Skin and subcutaneous tissue disorders) | 6 (7)
Right ear plugged (Ear and labyrinth disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Somnolence (General disorders) | 4 (4)
Sore throat (Gastrointestinal disorders) | 1 (1)
Strep throat (Infections and infestations) | 1 (1)
Thinning nails (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Tingling toes and feet (Nervous system disorders) | 2 (2)
Tingling, lips (Nervous system disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tooth abscess/infection (Gastrointestinal disorders) | 2 (2)
Tooth, cracked (General disorders) | 1 (1)
Tremor, upper extremity, hand (Nervous system disorders) | 3 (3)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Voice changes (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
Weakness (Nervous system disorders) | 3 (3)
Weakness, muscle (Musculoskeletal and connective tissue disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Xerostomia (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes